CLINICAL TRIAL: NCT03723148
Title: Compassionate Use of Fedratinib for Patients Who Have Previously Received TG101348, SAR302503 or Fedratinib
Brief Title: Individual Patient Compassionate Use of Fedratinib
Status: Available | Type: Expanded Access
Sponsor: Celgene (Industry)
Collaborators: Impact Biomedicines, Inc., a wholly owned subsidiary of Celgene Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: FEDR
Record Dates: First submitted 2018-10-25; First posted 2018-10-29 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Myelofibrosis
Keywords: Expanded Access; Compassionate Use
MeSH Terms: conditions — Primary Myelofibrosis | interventions — fedratinib

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Oral Fedratinib — Oral fedratinib administered as directed by treating physician.
  Other Names: FEDR

SUMMARY:
This is an expanded access program (EAP) for eligible participants designed to provide access to fedratinib.

Expanded access is only available in markets where fedratinib is not yet approved.

DETAILED DESCRIPTION:
This program is being offered on a patient by patient basis and will require company, Institutional Review Board/Independent Ethics Committee and Single Patient IND approval.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be considered if they received TG101348, SAR302503 or Fedratinib as a participant on a clinical trial prior to 31 Jan 2018.

Exclusion Criteria:

Subject is eligible for enrollment in an ongoing clinical trial using Fedratinib or has been treated with Fedratinib after 31 Jan 2018.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Celgene, Summit, New Jersey, United States